CLINICAL TRIAL: NCT03886740
Title: Tympanostomy Tubes Versus Eustachian Tube Dilation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty enrolling
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Hae-Ok Kim, Associate Professor of Otolaryngology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAS2555
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Eustachian Tube Dysfunction; Eustachian Tube Dysfunction of Left Ear; Eustachian Tube Dysfunction of Right Ear (Diagnosis); Eustachian Tube Dysfunction of Both Ears (Diagnosis)
Keywords: Eustachian Tube Dysfunction; Eustachian Tube balloon dilation; Eustachian Tube dilation; Tympanostomy
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: One arm will be treated with tympanostomy with pressure equalization tube placement and the other with Eustachian tube (ET) dilation. Their Eustachian Tube Dysfunction Questionnaire-7 scores will be collected over time and compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tympanostomy with tubes (Experimental): Tympanostomy with pressure equalization tube placement with Ventilation (Tympanostomy) Tubes
  Interventions: Procedure: Reducing symptoms of Eustachian tube dysfunction
- Eustachian tube (ET) dilation (Experimental): Eustachian tube (ET) dilation with ACCLARENT AERA® Eustachian Tube Balloon Dilation System
  Interventions: Procedure: Reducing symptoms of Eustachian tube dysfunction

INTERVENTIONS:
Procedure: Reducing symptoms of Eustachian tube dysfunction — One of two methods of reducing Eustachian Tube dysfunction will be performed and the Eustachian Tube Dysfunction Questionnaire-7 (ETDQ-7) scores will be compared

SUMMARY:
The objective of this study is to determine whether tympanostomy with pressure equalization tube placement or Eustachian tube (ET) dilation is superior at reducing symptoms of patients with ET dysfunction.

Given the apparent promise of Eustachian tube dilation and the lack of head to head comparison to the more traditional tympanostomy tube, this study seeks to compare them in a head to head manner in order to assess superiority in regards to ETDQ-7 and tympanogram improvements.

DETAILED DESCRIPTION:
The eustachian tube serves to ventilate and equalize middle ear pressure; clear secretions from the middle ear with mucociliary action; and protect the middle ear from sounds, pathogens, and secretions from the nasopharynx. First described anatomically by Eustachius in 1563 and with its exact function worked out a century later, Valsalva realized in 1703 that its opening was dynamic, not static, and described the namesake maneuver to expel pus from the middle ear into the external auditory canal. By the mid 18th century, multiple authors had attempted Eustachian tube catheterization and by the early 19th century, catheterization with irrigation and air insufflation had been described.(1) This shows how Eustachian tube dilation has been a known treatment for centuries, despite its relative obscurity prior to this decade. ET dysfunction is a common diagnosis many patients receiving care from an otologist or otolaryngologist receive. Dysfunction can be broken down into dilatory, which is caused by inflammation such as a virus, baro-challenge induced such as in scuba divers or those taking flights and patulous, which is of unclear etiology.(2) Symptoms are thought to include but are not limited to ear fullness, the sensation that the ear is underwater, otalgia, muffled hearing, tinnitus, autophony and ear popping amongst others. Clear diagnostic criteria are not present, though it is generally felt that a combination of symptoms and objective findings on otoscopy or tympanogram are enough to support the diagnosis. Many have resorted to using the Eustachian Tube Dysfunction Questionnaire-7 which is a validated symptom driven assessment, although it is only moderately associated with objective measures of ET dysfunction. (3,4) The only population-based study looking at prevalence used otoscopy, tympanogram and audiometry to estimate that it affects 0.9% of adults.(5) Unfortunately, there is currently no gold standard for treatment of ET dysfunction.

The only randomized control study of medical treatments showed no impact of nasal steroids on ET dysfunction.(6) The most common surgical option is a tympanostomy tube, which has been used since the 1950s for both middle ear effusions and ET dysfunction.(7) Tympanostomy tubes can alleviate tympanic membrane retraction, atelectasis and effusion, although they do not address the underlying etiology of the ET dysfunction. Numerous nonrandomized and or noncontrolled studies have showed improvement in symptoms with tympanostomy tube placement. Depending on the study and the definition, 70-100% improvement has been reported. Despite this, high-level evidence for tympanostomy tube efficacy in ET dysfunction remains lacking.(8) Adenoidectomy has also been proposed as a way to improve ET function, but not surprisingly, most studies have shown that it only helps if the adenoids are found to be abutting or obstructing the torus tubarii.(9,10) Furthermore, these studies focus on children, and the adenoid pad is not likely to be a contributing factor in most adults. Eustachian tube balloon dilation recently came back into the mainstream beginning with the 2010 study by Ockermann et al. which showed the procedure was safe and produced good results in a small cohort. Numerous studies since then have shown efficacy, including two separate multicenter randomized controlled trials published in 2017 and 2018. Both of these showed statistically and clinically significant superiority of ET balloon dilation over control as measured by improvement in ETDQ-7 and tympanogram type at up to 1 year. (11,12,13)

ELIGIBILITY:
Inclusion Criteria:

Determined to have chronic Eustachian tube dysfunction of at least 3 month duration based on a score of ≥ 14.5 on the Eustachian tube dysfunction questionnaire-7 (ETDQ-7), regardless of tympanogram status

Exclusion Criteria:

* Insurance that does reimburse for ET balloon dilation
* Patients with acute upper respiratory infection
* Tympanic membrane perforation
* Known middle ear disease such as cholesteatoma, acute otitits media, history of head and neck radiation, history of cleft palate, cystic fibrosis, ciliary dyskinesia, nasopharyngeal mass and patulous eustachian tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
ETDQ-7 score | Baseline
  The questionnaire contains 7 questions and total score will be divided by 7 to get mean score. Each visit will be averaged individually.
ETDQ-7 score | 6-weeks
  The questionnaire contains 7 questions and total score will be divided by 7 to get mean score. Each visit will be averaged individually.
ETDQ-7 score | 3-months
  The questionnaire contains 7 questions and total score will be divided by 7 to get mean score. Each visit will be averaged individually.
ETDQ-7 score | 6-months
  The questionnaire contains 7 questions and total score will be divided by 7 to get mean score. Each visit will be averaged individually.
ETDQ-7 score | 1-year
  The questionnaire contains 7 questions and total score will be divided by 7 to get mean score. Each visit will be averaged individually.
Tympanogram | Baseline
  The patient's post-op tympanogram will be recorded to compare to follow-up visits.
Tympanogram | 6-weeks
  The patient's post-op tympanogram will be compared to their pre-op tympanogram.
Tympanogram | 3-months
  The patient's post-op tympanogram will be compared to their pre-op tympanogram.
Tympanogram | 6-months
  The patient's post-op tympanogram will be compared to their pre-op tympanogram.
Tympanogram | 1 year
  The patient's post-op tympanogram will be compared to their pre-op tympanogram.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Kim, MD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feldmann H. [The Eustachian tube and its role in the history of otology. Images from the history of otorhinolaryngology, presented by instruments from the collection of the Ingolstadt German History Museum]. Laryngorhinootologie. 1996 Dec;75(12):783-92. doi: 10.1055/s-2007-997676. German. PMID 9081287
- [Background] Schilder AG, Bhutta MF, Butler CC, Holy C, Levine LH, Kvaerner KJ, Norman G, Pennings RJ, Poe D, Silvola JT, Sudhoff H, Lund VJ. Eustachian tube dysfunction: consensus statement on definition, types, clinical presentation and diagnosis. Clin Otolaryngol. 2015 Oct;40(5):407-11. doi: 10.1111/coa.12475. No abstract available. PMID 26347263
- [Background] McCoul ED, Anand VK, Christos PJ. Validating the clinical assessment of eustachian tube dysfunction: The Eustachian Tube Dysfunction Questionnaire (ETDQ-7). Laryngoscope. 2012 May;122(5):1137-41. doi: 10.1002/lary.23223. Epub 2012 Feb 28. PMID 22374681
- [Background] Teixeira MS, Swarts JD, Alper CM. Accuracy of the ETDQ-7 for Identifying Persons with Eustachian Tube Dysfunction. Otolaryngol Head Neck Surg. 2018 Jan;158(1):83-89. doi: 10.1177/0194599817731729. Epub 2017 Sep 26. PMID 28949806
- [Background] Browning GG, Gatehouse S. The prevalence of middle ear disease in the adult British population. Clin Otolaryngol Allied Sci. 1992 Aug;17(4):317-21. doi: 10.1111/j.1365-2273.1992.tb01004.x. PMID 1526050
- [Background] Gluth MB, McDonald DR, Weaver AL, Bauch CD, Beatty CW, Orvidas LJ. Management of eustachian tube dysfunction with nasal steroid spray: a prospective, randomized, placebo-controlled trial. Arch Otolaryngol Head Neck Surg. 2011 May;137(5):449-55. doi: 10.1001/archoto.2011.56. PMID 21576556
- [Background] Pappas JJ. Middle ear ventilation tubes. Laryngoscope. 1974 Jul;84(7):1098-117. doi: 10.1288/00005537-197407000-00004. No abstract available. PMID 4842776
- [Background] Llewellyn A, Norman G, Harden M, Coatesworth A, Kimberling D, Schilder A, McDaid C. Interventions for adult Eustachian tube dysfunction: a systematic review. Health Technol Assess. 2014 Jul;18(46):1-180, v-vi. doi: 10.3310/hta18460. PMID 25029951
- [Background] Nguyen LH, Manoukian JJ, Yoskovitch A, Al-Sebeih KH. Adenoidectomy: selection criteria for surgical cases of otitis media. Laryngoscope. 2004 May;114(5):863-6. doi: 10.1097/00005537-200405000-00014. PMID 15126745
- [Background] Bluestone CD, Cantekin EI, Beery QC. Certain effects of adenoidectomy of Eustachian tube ventilatory function. Laryngoscope. 1975 Jan;85(1):113-27. doi: 10.1288/00005537-197501000-00009. PMID 1089852
- [Background] Poe D, Anand V, Dean M, Roberts WH, Stolovitzky JP, Hoffmann K, Nachlas NE, Light JP, Widick MH, Sugrue JP, Elliott CL, Rosenberg SI, Guillory P, Brown N, Syms CA 3rd, Hilton CW, McElveen JT Jr, Singh A, Weiss RL Jr, Arriaga MA, Leopold JP. Balloon dilation of the eustachian tube for dilatory dysfunction: A randomized controlled trial. Laryngoscope. 2018 May;128(5):1200-1206. doi: 10.1002/lary.26827. Epub 2017 Sep 20. PMID 28940574
- [Background] Meyer TA, O'Malley EM, Schlosser RJ, Soler ZM, Cai J, Hoy MJ, Slater PW, Cutler JL, Simpson RJ, Clark MJ, Rizk HG, McRackan TR, D'Esposito CF, Nguyen SA. A Randomized Controlled Trial of Balloon Dilation as a Treatment for Persistent Eustachian Tube Dysfunction With 1-Year Follow-Up. Otol Neurotol. 2018 Aug;39(7):894-902. doi: 10.1097/MAO.0000000000001853. PMID 29912819
- [Background] Anand V, Poe D, Dean M, Roberts W, Stolovitzky P, Hoffmann K, Nachlas N, Light J, Widick M, Sugrue J, Elliott CL, Rosenberg S, Guillory P, Brown N, Syms C, Hilton C, McElveen J, Singh A, Weiss R, Arriaga M, Leopold J. Balloon Dilation of the Eustachian Tube: 12-Month Follow-up of the Randomized Controlled Trial Treatment Group. Otolaryngol Head Neck Surg. 2019 Apr;160(4):687-694. doi: 10.1177/0194599818821938. Epub 2019 Jan 8. PMID 30620688
- [Derived] Swords C, Smith ME, Patel A, Norman G, Llewellyn A, Tysome JR. Balloon dilatation of the Eustachian tube for obstructive Eustachian tube dysfunction in adults. Cochrane Database Syst Rev. 2025 Feb 26;2(2):CD013429. doi: 10.1002/14651858.CD013429.pub2. PMID 40008607